CLINICAL TRIAL: NCT02989610
Title: Post Market Clinical Follow Up Evaluating the Infinity Deep Brain Stimulation Implantable Pulse Generator System
Brief Title: Clinical Evaluation of the Infinity Deep Brain Stimulation System
Acronym: PROGRESS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10061
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: SJM-CIP-10061; PROGRESS; Infinity DBS; Parkinson Disease; UPDRS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Omnidirectional followed by directional DBS: Omnidirectional DBS is used for the first 3 months in all subjects, unless not tolerated. Directional DBS is used for months 3-6 in all subjects with a directional DBS lead. Primary end point is based on double-blind testing of omnidirectional vs. directional DBS in randomized order at 3-month follow-up visit.
  In this Observational study design, all interventions here are therapeutic interventions that are part of the standard of care, rather than assigned as part of an interventional study.
  Interventions: Device: Omnidirectional stimulation; Device: Directional stimulation

INTERVENTIONS:
Device: Omnidirectional stimulation — At the 3-month follow-up, therapeutic window, symptom relief and side effect thresholds are evaluated at the best level for omnidirectional stimulation with the Infinity DBS lead.
Device: Directional stimulation — At the 3-month follow-up, therapeutic window, symptom relief and side effect thresholds are evaluated using directional contacts at the best segmented level of the Infinity DBS lead.

SUMMARY:
The purpose of this post-market study is to characterize the clinical performance of the Infinity Deep Brain Stimulation (DBS) system, including the Implantable Pulse Generator (IPG), directional DBS leads, extensions, iPad clinician programmer, iPod patient controller and related system components.

Participants in the PROGRESS study are not assigned to interventional therapy groups. Participants in the PROGRESS study are followed in an observational format as they receive omnidirectional and then directional DBS programming that is part of routine medical care. Data on symptoms are collected during two different stages of programming, and those outcomes compared to assess the effect of omnidirectional or directional programming.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent;
* Subject is diagnosed with Parkinson's disease (PD) and has been recommended to receive an Infinity DBS system with a bilateral DBS implant in the Subthalamic Nucleus (STN), or has received an implant of an Infinity system with bilateral lead implants in the STN;
* Subject must be available for follow-up visits.

Exclusion Criteria:

* Subject is not a surgical candidate;
* In the investigator's opinion, the subject is unable to tolerate multiple programming sessions within a single setting;
* Subject is unable to comply with the follow-up schedule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have a diagnosis matching the approved indication and are being considered for a DBS implant or who have been implanted with an Infinity System comprise the target population for this study. All subjects who meet the inclusion and none of the exclusion criteria and have signed an Ethics Committee (EC) or Institutional Review Board (IRB) approved informed consent will be considered enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfons Schnitzler, MD, Principal Investigator — Heinrich-Heine-Universität Düsseldorf, Institute for Clinical Neuroscience; Jan Vesper, MD, Principal Investigator — Heinrich-Heine-Universität Düsseldorf, Department of Functional and Stereotactic Neurosurgery
Locations (41):
- United States (21):
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - Shands at University of Florida, Gainesville, Florida
  - University of Miami Hospital, Miami, Florida
  - Rush University, Department of Neurological Sciences, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - New York University Langone Medical Center - Tisch Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Medical, Columbus, Ohio
  - Oregon Health and Science University, Department of Neurology, Portland, Oregon
  - St. Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - Neurology Consultants of Dallas, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Abbott, Medical and Clinical Affairs, Plano, Texas
- Australia (3):
  - Princess Alexandra Hospital, Brisbane
  - Royal Melbourne Hospital - City Campus, Melbourne
  - Westmead Hospital, Richmond
- UZ Gent, Ghent, Belgium
- Germany (6):
  - Carl Gustav Carus Dresden an der Technischen, Dresden
  - Heinrich Heine University of Düsseldorf, Department of Neurology, Düsseldorf
  - Heinrich-Heine-Universität Düsseldorf, Department of Functional and Stereotactic Neurosurgery, Düsseldorf
  - UKE Hamburg, Hamburg
  - Johannes Gutenberg-University of Mainz, Mainz
  - Klinikum der Universität Regensburg, Regensburg
- Italy (3):
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia
  - Azienda Ospedaliero-Universitaria S Maria della Misericordia, Udine
- Poland (3):
  - Copernicus Hospital, Department of Neurosurgery,, Gdansk
  - Oncology Center- Marie Curie Institute, Warsaw
  - Institute of Psychiatry and Neurology, Warsaw
- Spain (3):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitario Central de Asturias, Department of Neurology,, Oviedo
  - Hospital Universitario Virgen del Rocío, Department of Neurology, Seville
- The Walton Centre, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, blinded-subject, blinded-evaluator, observational, multi-center 12-month post-market clinical follow-up study study enrolled a total of 234 participants between January 2017 and January 2019 at 37 sites in Europe, the U.S. and Australia. Of which 82 participants completed 36 months follow-up visit.
Groups:
- Omnidirectional Followed by Directional DBS: Omnidirectional DBS is used for the first 3 months in all subjects, unless not tolerated. Directional DBS is used for the following three months up to 6 months, unless not tolerated. At the three and twelve month follow-up visit therapeutic window, symptom relief and side effect thresholds are evaluated at the best level for omnidirectional and directional stimulation with the Infinity DBS lead.
Period: Overall Study
Arm/Group | Omnidirectional Followed by Directional DBS
Started | 234
Completed | 184
Not Completed | 50
Not completed — Withdrawal by Subject | 20
Not completed — Departure of PI from Site | 8
Not completed — Subject Participation Terminated by Investigator | 6
Not completed — Lost to Follow-up | 3
Not completed — Death | 3
Not completed — System Explant | 3
Not completed — Subject Non-Compliance | 2
Not completed — System Revision | 2
Not completed — PI Left, Study Closing | 1
Not completed — Site Discontinued Participation in the Study | 1
Not completed — Unable to Complete Visit Due to PI Leaving University | 1

BASELINE CHARACTERISTICS:
Arm/Group | Omnidirectional Followed by Directional DBS
Number analyzed (Participants) | 234
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 157
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 90
  Italy | 4
  Germany | 62
  Spain | 43
  Australia | 15
  Poland | 19
  Belgium | 1
Duration of Parkinson Symptoms [Mean (Standard Deviation); unit: Years] | 11.2 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With Wider Therapeutic Window With Directional Programming (Superiority)
Description: Therapeutic window is the range of stimulation amplitude that produces symptom relief without causing side effects. Proportion of subjects with a wider therapeutic window using directional stimulation, compared to a threshold of 60%. Based on randomized, double-blind evaluation using within-subject control.
Time Frame: 3-month follow-up visit after initial programming
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Omnidirectional Followed by Directional DBS
Number analyzed (Participants) | 204
Participants | 185
Statistical Analysis 1: Comparison: Omnidirectional Followed by Directional DBS; Proportion with wider therapeutic window using directional stimulation was compared to a performance goal of 60%; Test type: Superiority — Superiority hypothesis was that 95% lower confidence bound on proportion exceeded a threshold of 60%; p < 0.0001, Clopper-Pearson method

2. Secondary Outcome: Percentage Of Participants With Wider Therapeutic Window With Directional Programming (Non-Inferiority)
Description: Therapeutic window is the range of stimulation amplitude that produces symptom relief without causing side effects. The proportion of subjects with wider therapeutic window using directional stimulation will be compared to a performance goal of 60% with a non-inferiority threshold of 40%. Based on randomized, double-blind evaluation using within-subject control.
Time Frame: 3-month follow-up visit after initial programming
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Omnidirectional Followed by Directional DBS
Number analyzed (Participants) | 204
Participants | 185
Statistical Analysis 1: Comparison: Omnidirectional Followed by Directional DBS; Proportion with wider therapeutic window using directional stimulation was compared to a performance goal of 60%; Test type: Non-Inferiority — Non-inferiority hypothesis was that 95% lower confidence bound on proportion exceeded a threshold of 40%; p < 0.0001, Clopper-Pearson method

3. Secondary Outcome: Change In UPDRS III Score On and Off Stimulation (Medication On) at 3 and 6 Months
Description: Change with stimulation on vs. off in Unified Parkinson's Disease Rating Scale (UPDRS) part III motor examination at 3 months using omnidirectional stimulation, compared to 6 months using directional stimulation. UPDRS part III contains 27 questions used to measures severity of Parkinson's motor symptoms. The range of scores is 0 to 108, with higher score indicating greater symptoms. Subjects are on medication for the assessment.
Time Frame: 3 and 6 Months Follow-Up Visits
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Omnidirectional Followed by Directional DBS
Number analyzed (Participants) | 181
Score on a scale
  Omnidirectional stimulation (3 months) | 25.1 (12.8)
  Directional stimulation (6 months) | 30.8 (14.0)
Statistical Analysis 1: Comparison: Omnidirectional Followed by Directional DBS; Comparison of UPDRS part III on medication from 3 months using omnidirectional stimulation to 6 months using directional stimulation. The p-value presented is calculated and does not represent the threshold. The statistical test used for this endpoint is single sided, and the observed difference was in the opposite direction of the tested difference, leading to a p-value that is equivalent to 1 within the significance of the statistical software used; Test type: Superiority; p = 1.0000, t-test, 1 sided; Paired t-test

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | Omnidirectional Followed by Directional DBS
All-Cause Mortality (participants affected / at risk) | 3/234
Serious Adverse Events (participants affected / at risk) | 34/234
Other Adverse Events (participants affected / at risk) | 32/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omnidirectional Followed by Directional DBS (N=234)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1
Edema (Blood and lymphatic system disorders) | 1
Traumatic Psoas Bleed (Blood and lymphatic system disorders) | 1
Endocrinological Issues (Endocrine disorders) | 1
Appendicitis with Perforation (Gastrointestinal disorders) | 1
Umbilical Hernia (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Coma Related to Drowning (General disorders) | 1
Fall at Home (General disorders) | 1
Fracture of Vertebrae (General disorders) | 1
Several Falls (General disorders) | 1
Spinal Cord Canal Stenosis (General disorders) | 1
TLOC (Transient Loss of Consciousness) (General disorders) | 1
Sepsis Secondary to Influenza Infection (Infections and infestations) | 1
Battery Failure Within the Device (Injury, poisoning and procedural complications) | 2
Extension Fracture (Injury, poisoning and procedural complications) | 1
Lead Fracture (Injury, poisoning and procedural complications) | 1
Loss of Therapeutic Benefit - Change in Electrode Positions (Injury, poisoning and procedural complications) | 1
Speech or Language Impairment - Aphasia (Injury, poisoning and procedural complications) | 1
Speech or Language Impairment - Dysphagia (Injury, poisoning and procedural complications) | 1
Dystonia (Musculoskeletal and connective tissue disorders) | 1
Basal Cell Carcinoma of Scalp and Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Worsening of Motor/Parkinson's Disease Symptoms - Abnormal Gait (Nervous system disorders) | 1
Worsening of Motor/Parkinson's Disease Symptoms - Tremor (Nervous system disorders) | 1
Cognitive impairment - Confusion (Psychiatric disorders) | 1
Cognitive impairment - Disorientation (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dopamine Dysregulation Syndrome (Psychiatric disorders) | 1
Suicide (Psychiatric disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Renal Stones with Secondary Sepsis (Renal and urinary disorders) | 1
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Erosion (Skin and subcutaneous tissue disorders) | 1
Erosion Due to Undiagnosed Dermatologic Disorder (Skin and subcutaneous tissue disorders) | 1
Bioprosthetic Av Replacement (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omnidirectional Followed by Directional DBS (N=234)
Battery Failure Within the Device (Injury, poisoning and procedural complications) | 2
Cognitive Impairment - Depression (Psychiatric disorders) | 1
Cognitive Impairment - Emotional Lability (Psychiatric disorders) | 2
Cognitive Impairment - Hallucinations (Psychiatric disorders) | 1
Decreased Therapeutic Response (Injury, poisoning and procedural complications) | 2
Deep Brain Stimulation System Malfunction (Product Issues) | 1
Dyskinetic Dystonia (Musculoskeletal and connective tissue disorders) | 1
Dystonia (Musculoskeletal and connective tissue disorders) | 1
Headache/Migraine (General disorders) | 1
Impaired Wound Healing - Incision Site Drainage (Infections and infestations) | 1
Loss of Therapeutic Benefit - Change in Loose Electrical Connections (Injury, poisoning and procedural complications) | 1
Persistent Pain at Surgery Site or Ipg Site (Surgical and medical procedures) | 1
Sensory Disturbance or Impairment - Neuralgia (Nervous system disorders) | 1
Sensory Disturbance or Impairment - Sensory Deficit (Injury, poisoning and procedural complications) | 2
Shortness of Breath On Exertion (Respiratory, thoracic and mediastinal disorders) | 1
Skull Discoloration (Injury, poisoning and procedural complications) | 1
Speech or Language Impairment - Dysarthria (Injury, poisoning and procedural complications) | 1
Sub-Optimal Placement of Lead (Injury, poisoning and procedural complications) | 1
Undesirable Changes in Stimulation - Other (Injury, poisoning and procedural complications) | 2
Worsening of Motor/Parkinson's Disease Symptoms - Abnormal Gait (Nervous system disorders) | 2
Worsening of Motor/Parkinson's Disease Symptoms - Bradykinesia (Nervous system disorders) | 2
Worsening of Motor/Parkinson's Disease Symptoms - Dyskinesia (Nervous system disorders) | 7
Worsening of Motor/Parkinson's Disease Symptoms - Motor Fluctuations (Nervous system disorders) | 1
Worsening of Motor/Parkinson's Disease Symptoms - Rigidity (Nervous system disorders) | 1
Worsening of Motor/Parkinson's Disease Symptoms - Tremor (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT02989610/Prot_SAP_001.pdf